CLINICAL TRIAL: NCT00989716
Title: A Prospective, Collaborative, International, Multicentre, Randomised, Parallel-group, Single and Outcome Blinded, Controlled, Factorial Trial to Investigate the Safety and Efficacy of Treatment With Transdermal Glyceryl Trinitrate, a Nitric Oxide Donor, and of Continuing or Stopping Temporarily Pre-stroke Antihypertensive Therapy, in Patients With Acute Stroke
Brief Title: The Efficacy of Nitric Oxide in Stroke (ENOS) Trial
Acronym: ENOS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 04002; ISRCTN99414122; EudraCT no: 2004-003870-27
Record Dates: First submitted 2009-10-02; First posted 2009-10-05 (Estimated); Last update posted 2012-07-24 (Estimated); Status verified 2012-07

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Glyceryl trinitrate transdermal patch (Active Comparator)
  Interventions: Drug: Transdermal glyceryl trinitrate patch
- Continue or stop pre-stroke antihypertensives (Experimental)
  Interventions: Drug: Pre-stroke antihypertensives

INTERVENTIONS:
Drug: Transdermal glyceryl trinitrate patch — 5mg per day
  Other Names: Local ward stock to be used.
  Arms: Glyceryl trinitrate transdermal patch
Drug: Pre-stroke antihypertensives — Continue or stop pre-stroke anti-hypertensives
  Arms: Continue or stop pre-stroke antihypertensives

SUMMARY:
Nitric oxide is a multimodal candidate treatment for acute stroke having a number of properties which may be beneficial in acute stroke, including lowering blood pressure, causing cerebral vasodilation, and improving central and systemic haemodynamics. Nitric oxide donors are effective in experimental stroke and pilot studies in patients suggest that one, glyceryl trinitrate, can be delivered easily in a transdermal preparation. Around half of all patients admitted with acute stroke are taking antihypertensive therapy immediately prior to their stroke. No data exist as to whether it is beneficial or safe to stop or continue this treatment during the acute phase. ENOS is a prospective, international, multicentre, randomised, parallel-group, blinded, controlled, collaborative, factorial trial designed to test two questions related to the management of blood pressure immediately post-stroke:

1. The safety and efficacy of nitric oxide, given as transdermal glyceryl trinitrate.
2. The safety and efficacy of stopping or continuing prior antihypertensive medication.

Previously independent adult patients who are conscious and have residual limb weakness are eligible for enrollment. Central randomisation will be performed via the internet. Treatment is initiated within 48 hours of stroke onset and is given as daily glyceryl trinitrate patches for 7 days. A computed tomography (CT) scan is required within 7 days of randomisation. Early follow-up is performed locally over the 7 days of treatment, including blood pressure, early stroke events, and adverse events. Telephone central follow-up by the trial co-ordinating centre will be performed at 3 months. The primary outcome is combined death or dependency (modified Rankin Score >2).

ELIGIBILITY:
Inclusion Criteria:

* Adult(> 18 yrs).
* Clinical stroke syndrome with limb weakness lasting at least 1 hour i.e. not likely to be a transient ischaemic attack).
* Limb weakness (SNSS Arm <6 and/or Leg <6).
* Onset < 48 hours.
* Conscious (Glasgow Coma Scale > 8).
* Independent prior to stroke (pre-morbid Rankin scale < 2).
* Meaningful consent, or assent from a relative or carer

Exclusion Criteria:

* Definite need for nitrate therapy
* Contraindication to nitrate therapy
* Definite need for prior antihypertensive or anti-anginal medication
* Definite need for antihypertensive therapy during acute stroke
* Systolic blood pressure <140 mmHg or >220 mmHg.
* Patients expected to require surgical intervention
* Known intracerebral pathology other than stroke
* Other serious condition which is likely to prevent outcome assessment at 3 months
* Previous enrollment in ENOS or current involvement in another trial of an experimental drug intervention.
* Not available for follow-up -Females of childbearing potential, pregnancy or breastfeeding. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3500 (Estimated)
Dates: Start 2001-07; Primary Completion 2013-10 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Reduced death or dependency (modified Rankin score) | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Philip Bath, Principal Investigator — University of Nottingham
Locations (1):
- Nottingham University Hospitals NHS Trust (City Hospital), Nottingham, Nottinghamshire, United Kingdom

REFERENCES:
- [Derived] Learoyd AE, Woodhouse L, Shaw L, Sprigg N, Bereczki D, Berge E, Caso V, Christensen H, Collins R, Czlonkowska A, El Etribi A, Farr TD, Gommans J, Laska AC, Ntaios G, Ozturk S, Pocock SJ, Prasad K, Wardlaw JM, Fone KC, Bath PM, Trueman RC; ENOS Trial investigators. Infections Up to 76 Days After Stroke Increase Disability and Death. Transl Stroke Res. 2017 Dec;8(6):541-548. doi: 10.1007/s12975-017-0553-3. Epub 2017 Jul 27. PMID 28752410
- [Derived] Woodhouse L, Scutt P, Krishnan K, Berge E, Gommans J, Ntaios G, Wardlaw J, Sprigg N, Bath PM; ENOS Investigators. Effect of Hyperacute Administration (Within 6 Hours) of Transdermal Glyceryl Trinitrate, a Nitric Oxide Donor, on Outcome After Stroke: Subgroup Analysis of the Efficacy of Nitric Oxide in Stroke (ENOS) Trial. Stroke. 2015 Nov;46(11):3194-201. doi: 10.1161/STROKEAHA.115.009647. Epub 2015 Oct 13. PMID 26463698
- See also: Related Info — http://www.enos.ac.uk